CLINICAL TRIAL: NCT02962596
Title: European Multicenter Validation of an ADNEXMR SCORING System for Characterizing Adnexal Masses: EURAD-MR Classification
Brief Title: EURAD MRI Classification of US Indeterminate Adnexa Lesions
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: 2014-0112; A539320 (Other: UW Madison); SMPH/RADIOLOGY/RADIOLOGY (Other: UW Madison)
Record Dates: First submitted 2016-10-31; First posted 2016-11-11 (Estimated); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Ovarian Tumor
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: ADNEXMR SCORING system — Scoring system used to standardize the imaging report for sonographically indeterminate adnexal masses.

SUMMARY:
This research is targeting patients with sonographically indeterminate adnexal mass that are being referred for clinical MR imaging. Investigators from the UW will be contributing coded MR images and associated health information (US results, laboratory/pathology results) to the EURAD trial. In addition, outcomes data on each patient will be sent at month 24 of the research.

DETAILED DESCRIPTION:
An adnexal mass is the most common indication for gynaecological surgery. Pre operative characterization is crucial and a scoring system would be useful to standardize the imaging report and thus, improve patients management. Recently, the coordinating center developed the first MR scoring system named ANDEXMR SCORING system in a retrospective study which is accurate and reproducible. The objectives of this trial are to perform an external prospective validation of this scoring system to evaluate its potential impact on therapeutic strategy and to test its reproducibility.

This is a prospective large multicenter study. All patients with a sonographically indeterminate adnexal mass referred for MR imaging will be included from each participating center. One senior and one junior radiologists independently analyze the different MR criteria to characterize adnexal masses. The reader will then classify the mass using ADNEXMR SCORING system.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years of age or older
* With indeterminate ultrasonographic adnexal mass

Exclusion Criteria:

* Patients under 18 years of age

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with an indeterminate ultrasonographically adnexal mass referred for MR imaging
Sampling Method: Non-Probability Sample
Enrollment: 1340 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-10-14 (Actual); Study Completion 2018-08-15 (Actual)

PRIMARY OUTCOMES:
Reproducibility of the ADNEX MR scoring system between centers | 24 months
  Evaluate if ADNEXMR SCORING system is relevant for reporting pelvic magnetic resonance imaging (MRI) examinations performed for characterization of sonographically indeterminate adnexal masses in an external prospective multicenter study

SECONDARY OUTCOMES:
Differences in rate of surgery in women with adnexal lesions in those where the ADNEX MR score is used compared to when it is not used. | 24 months
  The potential impact of applying the score to the therapeutic strategy, in particular to measure the possible reduction in unnecessary surgery in benign cases.
Reproducibility of the score | 24 months
  If ADNEXMR SCORING system improves reproducibility of MR report for characterization of adnexal masses
Comparison between a blinded and an unblinded radiologist regarding sonographic data | 24 months
  If ADNEXMR SCORING system is as accurate if the radiologist is blinded from any clinical and ultrasonographic data

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Sadowski, MD, Principal Investigator — University of Wisconsin, Madison; Isabelle Thomassin-Naggara, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Andrea Rockall, MD, Study Director — Imperial College of London
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Images and associated data will be labeled with a unique study number that identifies the research site and the patient number (e.g. UWisc001). The link to identifiable information will remain at the University of Wisconsin

REFERENCES:
- [Result] Thomassin-Naggara I, Poncelet E, Jalaguier-Coudray A, Guerra A, Fournier LS, Stojanovic S, Millet I, Bharwani N, Juhan V, Cunha TM, Masselli G, Balleyguier C, Malhaire C, Perrot NF, Sadowski EA, Bazot M, Taourel P, Porcher R, Darai E, Reinhold C, Rockall AG. Ovarian-Adnexal Reporting Data System Magnetic Resonance Imaging (O-RADS MRI) Score for Risk Stratification of Sonographically Indeterminate Adnexal Masses. JAMA Netw Open. 2020 Jan 3;3(1):e1919896. doi: 10.1001/jamanetworkopen.2019.19896. PMID 31977064